CLINICAL TRIAL: NCT07239011
Title: Dapagliflozin, an SGLT2 Inhibitor, From Oral Hypoglycemic Agent to Antidepressant Drug
Brief Title: Dapagliflozin in Depression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8759
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group (n =30) who will receive fluoxetine (20 mg) and placebo once daily for 3 months
  Interventions: Drug: Fluoxetine
- Dapagliflozin group (Active Comparator): Dapagliflozin group (n=30) who will receive fluoxetine (20 mg) once daily plus dapagliflozin 10 mg once daily for 3 months
  Interventions: Drug: Fluoxetine; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine is an antidepressant medication of the selective serotonin reuptake inhibitor class used for the treatment of major depressive disorder, anxiety, obsessive-compulsive disorder, panic disorder, premenstrual dysphoric disorder, and bulimia nervosa.
Drug: Dapagliflozin — Dapagliflozin is a medication used to treat type 2 diabetes. It is also used to treat adults with heart failure and chronic kidney disease. It reversibly inhibits sodium-glucose co-transporter 2 (SGLT-2) in the renal proximal convoluted tubule to reduce glucose reabsorption and increase urinary glucose excretion.
  Arms: Dapagliflozin group

SUMMARY:
Major depressive disorder (MDD) is currently one of the leading causes of disability and suicidal death worldwide, and despite extensive research and massive improvements in mental health, the nature of MDD remains ambiguous. Moreover, about two-thirds of MDD patients fail to optimally respond to currently available standard therapies, and many of them suffer from treatment-resistant depression

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Both male and female will be included Negative pregnancy test and effective contraception. Depressed patients for at least 2 months with Hamilton rating score more than 18.

Exclusion Criteria:

Patients with bipolar I or bipolar II disorder, personality disorders, and eating disorders.

Patients with substance dependence or abuse Patients with history of seizures or receiving electroconvulsive therapy (ECT) Patients with inflammatory disorders Patients with allergy or contraindications to the used medications Patients with finally pregnant or lactating females Diabetic patients Sever kidney disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure was the 17-item HDRS. | 3 months
  All patients will be assessed via Hamilton Depression Rating Scale (HDRS). A HDRS score of ≤ 7 indicates remission or partial remission [HDRS<17 and>7]. Response was defined as ≥ 50% drop in the HDRS score.

SECONDARY OUTCOMES:
Change in quality of life. | 3 months
  Change in quality of life will be assessed through Short Form-36 Health Survey. One of the most commonly used quality of life tools. It consists of 36 items, and 8 domains

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt